CLINICAL TRIAL: NCT03707496
Title: A Registry of De Winter Symdrome of Hainan General Hospital
Brief Title: A Registry of De Winter Symdrome of Single Center
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hainan People's Hospital (Other)
Responsible Party: Principal Investigator, Liao Wang, Principal Investigator, Hainan People's Hospital
Other Study IDs: Reg001
Record Dates: First submitted 2018-10-08; First posted 2018-10-16 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: ACS - Acute Coronary Syndrome
Keywords: De Winter Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DeWinterCohort: Patients with de Winter syndrome pattern ECG

SUMMARY:
This registry started January 1,2018 to collect patients who diagnosed as De Winter Symdrome for the first time in Hainan General Hospital.All enrolled patients will receive 30 days followed-up.

ELIGIBILITY:
Inclusion Criteria:

* Index ECG ST segment showed a 1- to 3-mm upsloping ST-segment depression at the J point in leads V1 to V6 that continued into tall, positive symmetrical T waves
* Received coronary angiography during hospitalization

Exclusion Criteria:

-No coronary angiography results was available during hospitalization

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All acute coronary syndrome patients with a de Winter syndrome ECG pattern
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with MACEs within 30 days | 30 days
  Number of participants with cardiac death,non-fatal myocardial infarction,stroke,heart failure in 30 days

SECONDARY OUTCOMES:
Number of participants with MACEs In-hospital | throughout current hospitalization
  Number of participants with cardiac death,non-fatal myocardial infarction,stroke,heart failure in-hospital
Number of Participants with MACEs within 7 days after admitted | 7 days after admitted
  Number of participants with cardiac death,non-fatal myocardial infarction,stroke,heart failure in 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hainan General Hospital, Haikou, Hainan, China